CLINICAL TRIAL: NCT05690672
Title: Screening for Delirium in Older Inpatients Using 3D-CAM and 4AT: Protocol for a Randomized Pilot Study
Brief Title: Screening for Delirium in Older Inpatients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Johannes Riis Jensen, Principal Investigator, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: N-20220026
Record Dates: First submitted 2022-09-26; First posted 2023-01-19 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Delirium in Old Age

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D-CAM screening (Active Comparator)
  Interventions: Diagnostic Test: Delirium Screening
- 4AT screening (Active Comparator)
  Interventions: Diagnostic Test: Delirium Screening

INTERVENTIONS:
Diagnostic Test: Delirium Screening — Either 3D-CAM or 4AT

SUMMARY:
Two-arm parallel-randomized pilot study and to collect data at the Department of Geriatric Medicine at Aalborg University Hospital. The aim is to assess the feasibility of a future randomized controlled study comparing Danish versions of 3D-CAM and 4AT in an acute medical setting. The primary objective is to assess 1) feasibility of obtaining informed consent and recruiting older adults within 24 hours of admission (or surgery) at the Department of Geriatric Medicine, Department of Acute Medicine, or Department of Orthopedic Surgery. Secondary objectives are 2a) to compare feasibility of recruitment and testing in the three different departments, 2b) to inform a preliminary evaluation of validity and reliability of the Danish version of screening instruments, and 2c) to obtain data on variance to support calculating sample size for a full-scale RCT.

DETAILED DESCRIPTION:
We will recruit participants through a consecutive sampling of all potentially eligible patients. Recruitment will take place in three different settings: the Department of Geriatric Medicine, the Department of Acute Medicine, and the Department of Orthopedic Surgery. One week will be allocated for recruitment in each setting.

Potentially delirious patients often have impaired cognitive status. Therefore, the process of recruitment and informed consent is critically important and poses a central issue of feasibility to be assessed in this study.

It cannot be known with certainty whether patients are delirious prior to inclusion into the study, and even among delirious patients, there are considerable circadian fluctuations (as this is a hallmark of the condition), meaning that patients may have lucid moments during the day where they are cognitively intact and may be able to give informed consent.

Generally, informed consent will be sought from participants when possible. In case they are permanently or temporarily unable to give informed consent, informed consent will be sought from next of kin. Due to the short time in the study for each participant, it is not anticipated that participants will regain the ability to give informed consent during the study. However, if they do, new informed consent will be obtained from the participant. The number of potential participants at each step will be documented to assess problems with feasibility.

ELIGIBILITY:
Inclusion Criteria:

* Age over 80 years
* Admission or surgery within the last 24 hours

Exclusion Criteria:

* Unable to obtain contact to next of kin for informed consent within time-frame

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-09-28 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruitment overall | 3 weeks total
  Measured by counting the number of participants giving informed consent, as well as number of participants in each setting not giving informed consent in each setting over the 3 week period.

SECONDARY OUTCOMES:
Feasibility of recruitment in different settings | 1 week each
  Comparison of the number of participants (counted) recruited in the Department of Orthopedic Surgery, Geriatric Medicine and Acute Medicine
Validity of screening tools | 3 weeks total
  Preliminary results of screening validity of 4A's test and 3D-CAM test comparing sensitivity and specificity

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University Hospital, Aalborg, Northern Jutland, Denmark